CLINICAL TRIAL: NCT04595175
Title: Changes in Seroprevalence and Wellness Over Time in Healthcare Workers (CONSERVE-HCW)
Acronym: CONSERVE-HCW
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brian Tiffany, MD (Other)
Collaborators: Chandler Regional Medical Center (Unknown); Arizona General Hospital (Unknown); Mercy Gilbert Medical Center (Unknown)
Responsible Party: Sponsor-Investigator, Brian Tiffany, MD, Chief Medical Officer, St. Joseph's Hospital and Medical Center, Phoenix
Organization: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Other Study IDs: 20-510-157-66-21
Record Dates: First submitted 2020-06-10; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: COVID-19 Infection
Keywords: Serology; Wellness; SARS-CoV-2 IgG; Seroprevalence; Healthcare Workers
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — One tube of blood will be sent to the appropriate hospital lab for the Abbott IgG testing. The other two tubes of blood will be processed and biobanked. The same tubes will be drawn on the subsequent visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Investigators propose a multi-center, observational, longitudinal, cohort study of the serology and wellness of HCWs over a year of the COVID-19 pandemic.

DETAILED DESCRIPTION:
All consenting participants will undergo survey assessment and diagnostic testing with the Abbott Architect SARS-CoV-2 IgG assay (IgG) every three months for a one year period. Clinical outcomes and related data capture will be performed at this same interval.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years; and
2. Be an active member of the CommonSpirit Health workforce or medical staff during the COVID-19 pandemic and at the time of enrollment; and
3. Have access to the Internet; and
4. The ability to provide informed consent.

Exclusion Criteria:

1. Subjects that lack the ability for longitudinal follow-up; and/or
2. Subjects that do not meet the above inclusion criteria. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be enrolled across CommonSpirit Health hospitals and care facilities (all branded as Dignity Health) at five sites in Maricopa County, Arizona: Arizona General Hospital, Chandler Regional Medical Center, Mercy Gilbert Medical Center, St. Joseph's Hospital and Medical Center and St. Joseph's Westgate Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Baseline IgG Assay Information | Baseline
  Seroprevalence of anti-SARS-CoV-2 IgG antibodies in HCWs
Change in IgG Assay Information | From Baseline to 3 months, 6 months, 9 months, & 12 months
  The change in the seroprevalence of anti-SARS-CoV-2 IgG antibodies in HCWs over one year.
Compare seroprevalence of anti-SARS-CoV-2 IgG antibodies between groups | From Baseline to 3 months, 6 months, 9 months, & 12 months
  Compare seroprevalence of anti-SARS-CoV-2 IgG antibodies in 'front-line' workers and non-'front-line' HCWs
Impact of COVID-19 Pandemic on Perceived Wellness and Job Satisfaction | Baseline to 12 months
  Over the 12 months of the study, evaluate the impact of the COVID-19 pandemic on HCW wellness using the Perceived Wellness Survey. Job satisfaction will be measured using a locally developed questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Tiffany, MD, PhD, Principal Investigator — Chief Medical Officer Dignity Health Arizona
Locations (1):
- Chandler Regional Medical Center, Chandler, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- See also: COVID-19 Death toll — https://globalnews.ca/news/6729174/coronavirus-spain-death-toll-china/
- See also: Healthcare worker COVID-19 infection rates — https://www.cebm.net/covid-19/covid-19-how-many-healthcare-workers-are-infected/